CLINICAL TRIAL: NCT00623337
Title: Cluster Randomised Trial to Evaluate the Impact of Routine Home Visits to Provide a Package of Essential Newborn Care Interventions in the Third Trimester of Pregnancy and the 1st Week of Life on Neonatal Mortality in Rural Ghana
Brief Title: Ghana Newborn Home Visits Neonatal Mortality Trial
Acronym: Newhints
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Newhints; WHO: C6-181-512,# 007; SNL: Sub-grant # 251; LSHTM: EPNPVE28 & EPNPVP18
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2010-02

CONDITIONS: Neonatal Mortality
Keywords: care seeking; pregnancy and childbirth; newborn care practices; low birth weight babies
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Newhints (Experimental): Home visits
  Interventions: Behavioral: Home visits
- Control (No Intervention): Community based surveillance volunteers will continue with current duties eg urging attendance at immunisation clinics and child health weeks

INTERVENTIONS:
Behavioral: Home visits — Home visits by community based surveillance volunteers (2 during pregnancy & 3 during 1st week of life) to promote facility delivery, careseeking during pregnancy and childbirth and essential newborn care practices and to identify & refer sick babies
  Arms: Newhints

SUMMARY:
Introduction: Just under four million infants die each year before reaching one month of age; neonatal deaths now account for 38% of the 10.8 million deaths among children younger than 5 years of age. Tackling neonatal mortality is essential if the millennium development goal to reduce by 2015 overall child mortality by two-thirds from its levels in 1990 is to be achieved. Postnatal care for mothers and neonates in developing countries, particularly when deliveries occur at home, is either not available or is of poor quality. Trained community workers are considered by many to be pivotal to newborn care in the community, as they can act as catalysts for community actions and also be providers of care.Reductions in neonatal mortality have been slower in Sub-Saharan Africa than in any other region, and no evaluations of the effectiveness and feasibility of home visits in reducing neonatal mortality have been conducted.

Trial aim: To link with the Ghana Health Service to develop a feasible and sustainable intervention to improve newborn care practices and careseeking during pregnancy and childbirth, and to identify and refer very low birth weight and/or sick babies, through routine home-visits by community health workers (CHWs), and by so doing reduce neonatal mortality.

DETAILED DESCRIPTION:
Study area: The NEWHINTS trial will be conducted in 6 contiguous districts with an area of 12,000km in the central Brong Ahafo Region of rural Ghana. The area is predominantly rural and has a total population of approximately 600,000 persons, with more than 100,000 women of reproductive age. The study area is multi-ethnic and education levels are low. It is served by 4 district hospitals, and a small number of additional government health centres and private facilities. More than 15,000 babies are born within the area each year; the neonatal mortality rate is about 30 per 1000 live births. Over 50% of births occur at home and these home deliveries account for a large proportion of all neonatal deaths. A potential cadre of CHWs, who are currently working in the region and whose capacity could be expanded to include home visits, are Community Based Surveillance Volunteers (CBSVs); CBSVs currently assist the DHMTs with the registration of births, disease detection and community mobilization.

Intervention: The intervention is being developed by a collaborative group from Kintampo Health Research Centre, the District Health Management Teams (DHMTs) of the 6 districts and the London School of Hygiene and Tropical Medicine. It will comprise of:

1. Training CBSVs to identify pregnant women in the community and to conduct 2 home visits during pregnancy and 3 in the first week of life of the infant on days 1, 3 and 7:

   * to promote birth preparedness and prompt careseeking during pregnancy and childbirth
   * to promote essential perinatal and neonatal care practices
   * to identify and refer very low birth weight or sick babies
   * to give advice on special treatment for low birth weight babies
   * to teach neonatal danger signs and encourage prompt careseeking
   * to promote key child survival interventions for infancy (breastfeeding, bednets, immunisations) CBSVs will provide support through dialogue and problem-solving. Other family members key in decision-making concerning childbirth and newborn care will be invited to take part in the discussions.
2. Developing a sustainable supervisory and remuneration structure for the CBSVs;
3. Various intervention support activities inc

   * Sensitisation of health facility staff to intervention messages and approach#
   * Sensitisation of traditional birth attendants (TBAs)
   * Meetings with village leaders to introduce intervention aims and activities
   * Community durbars

Study design: Formative research consisting of in-depth interviews, focus-groups and pilot trials of home visits/improved practices will be conducted to improve the feasibility and optimality of the planned intervention and to design training and intervention support materials. A cluster randomised controlled trial design with 98 health zones as units of randomisation will be used to evaluate the impact on neonatal mortality, careseeking during pregnancy and childbirth and newborn care practices. The intervention will be implemented in half of the zones, chosen at random, and evaluated over an 18 month period. Impact data will come from ongoing 4-weekly surveillance of all women of child-bearing age and their infants including verbal post mortems, conducted as part of the ongoing "ObaapaVitA" Vitamin A and maternal mortality trial. A process evaluation will be conducted over 3-monthly intervals to assess the coverage and quality of the services provided and the response to the services.

ELIGIBILITY:
Inclusion Criteria:

* All live births in trial area

Exclusion Criteria:

* None

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15000 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality rate | deaths within 28 days of birth

SECONDARY OUTCOMES:
% mothers carrying out promoted newborn care practices | within 28 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Betty R Kirkwood, Principal Investigator — London School of Hygiene and Tropical Medicine; Zelee E Hill, Principal Investigator — Institute of Child Health, London; Alexander Manu, Principal Investigator — Kintampo Health Research Centre (KHRC); Charlotte Tawiah, Principal Investigator — KHRC; Seth Owusu-Agyei, Principal Investigator — KHRC
Locations (1):
- Kintampo Health Research Centre, Kintampo, Brong Ahafo Region, Ghana

REFERENCES:
- [Background] Hill Z, Manu A, Tawiah-Agyemang C, Gyan T, Turner K, Weobong B, Ten Asbroek AH, Kirkwood BR. How did formative research inform the development of a home-based neonatal care intervention in rural Ghana? J Perinatol. 2008 Dec;28 Suppl 2:S38-45. doi: 10.1038/jp.2008.172. PMID 19057567
- [Derived] Lohela TJ, Nesbitt RC, Manu A, Vesel L, Okyere E, Kirkwood B, Gabrysch S. Competence of health workers in emergency obstetric care: an assessment using clinical vignettes in Brong Ahafo region, Ghana. BMJ Open. 2016 Jun 13;6(6):e010963. doi: 10.1136/bmjopen-2015-010963. PMID 27297010
- [Derived] Manu A, Hill Z, Ten Asbroek AH, Soremekun S, Weobong B, Gyan T, Tawiah-Agyemang C, Danso S, Amenga-Etego S, Owusu-Agyei S, Kirkwood BR. Increasing access to care for sick newborns: evidence from the Ghana Newhints cluster-randomised controlled trial. BMJ Open. 2016 Jun 13;6(6):e008107. doi: 10.1136/bmjopen-2015-008107. PMID 27297006
- [Derived] Vesel L, Manu A, Lohela TJ, Gabrysch S, Okyere E, Ten Asbroek AH, Hill Z, Agyemang CT, Owusu-Agyei S, Kirkwood BR. Quality of newborn care: a health facility assessment in rural Ghana using survey, vignette and surveillance data. BMJ Open. 2013 May 9;3(5):e002326. doi: 10.1136/bmjopen-2012-002326. PMID 23667161
- [Derived] Kirkwood BR, Manu A, ten Asbroek AH, Soremekun S, Weobong B, Gyan T, Danso S, Amenga-Etego S, Tawiah-Agyemang C, Owusu-Agyei S, Hill Z. Effect of the Newhints home-visits intervention on neonatal mortality rate and care practices in Ghana: a cluster randomised controlled trial. Lancet. 2013 Jun 22;381(9884):2184-92. doi: 10.1016/S0140-6736(13)60095-1. Epub 2013 Apr 9. PMID 23578528
- [Derived] Kirkwood BR, Manu A, Tawiah-Agyemang C, ten Asbroek G, Gyan T, Weobong B, Lewandowski RE, Soremekun S, Danso S, Pitt C, Hanson K, Owusu-Agyei S, Hill Z. NEWHINTS cluster randomised trial to evaluate the impact on neonatal mortality in rural Ghana of routine home visits to provide a package of essential newborn care interventions in the third trimester of pregnancy and the first week of life: trial protocol. Trials. 2010 May 17;11:58. doi: 10.1186/1745-6215-11-58. PMID 20478070